CLINICAL TRIAL: NCT05477420
Title: A Survey Study and Effect of Web-based Decision Aids on Preferences Shift
Brief Title: Effect of Web-based Decision Aids on Preferences Shift
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Winnie W.S. MAK, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SBRE- 20-275
Record Dates: First submitted 2022-07-06; First posted 2022-07-28 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Depression; Psychotherapies
Keywords: Depression; Online psychotherapies; psychotherapies; Decision aid
MeSH Terms: conditions — Depression | interventions — Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Participants in the experimental group will be expected use the decision aid developed in this study. They will be assessed at two different time points:
  (1) before intervention (T0) and (2) post-intervention (T1).
  Interventions: Other: Decision Aid
- Attention control group (No Intervention): The control group participants will be asked to search information related to "Depression" and "therapies for Depression" online. They will be assessed at two different time points:
  (1) at baseline (T0) and (2) after searching for information (T1).

INTERVENTIONS:
Other: Decision Aid — Participants in the experimental group would be asked to use the decision aid developed by the study. The decision aid tool will ask participants their preferences on traditional face-to-face and online psychotherapies and how they rank different treatment attributes.
  Arms: Experimental group

SUMMARY:
The goals of this study is to examine whether treatment preferences shift after receiving a clients' decision aids about psychotherapy in digital and in in-person format.

DETAILED DESCRIPTION:
1.1 The importance of clients' Preference and Acceptability While introducing and implementing E-mental health service, clients' preference and acceptability should not be neglected. It is increasingly acknowledged that acceptability should be considered when designing, evaluating, and implementing novel healthcare interventions. Treatment acceptability has also been framed as a key factor for successful dissemination and implementation of any new health service model, because A given treatment may be clinically effective, yet unacceptable for clients and patients(Kaltenthaler et al., 2008; Wallin, Mattsson, &Olsson, 2016). Besides, clients' preference and acceptability of may not merely influence satisfaction, but also have significant implications for adherence and outcome (Gelhorn, Sexton, &Classi, 2011). For example, according to a meta-analytic review across various treatment formats, individuals who matched with preferred treatment had a higher chance of showing improvements and were almost half as likely to drop out of treatment compared to those whose preferred choice of treatment were not offered(Swift &Callahan, 2009). Previous studies also suggested that preferences and acceptability are significantly related to important process and outcomes of treatment such as service initiation, adherence, compliance, engagement, and the development of working alliance (Gelhorn et al., 2011). Thus, not only did the German National Care Guideline (S-3-Guideline, 2nd edition) for unipolar depression recommends a seven-step model of shared decision-making for health care service institutes and demands that the assessment and consideration of client preferences should be an indispensable step within the decision making process(German Medical Association, 2015). This year NICE has also published new guidelines recommending shared decision making be part of everyday practice across all healthcare settings(National Institute for Clinical Excellence, 2021).

Nevertheless, in the field of E-mental health for depression, studies investigating treatment preferences are not abundant and have predominantly focused on contrasting the choice between psychotherapy and pharmacological therapy (Raue, Schulberg, Heo, Klimstra, &Bruce, 2009; Steidtmann et al., 2012). The homogenous scope of studies leaves new treatment modality like the use of technology aside, although there were still a handful of articles on this topic. For example, Renn et. al (2019) found that 44.5% of participants preferred in-person psychotherapy and 25.6% preferred self-guided digital treatment; March et. al (2018) found a significant proportion of respondents (39.6%) endorsed intentions to use e-mental health services if experiencing mental health difficulties in the future; yet Musiat, Goldstone, &Tarrier (2014) reported a low likelihood of using computerized treatments for mental health in the future, and contrarily McCall, Sison, Burnett, Beahm, &Hadjistavropoulos (2020) found that vast majority of participants (93%) reported that they would access E-mental health service if they needed help with mental health problems. Although most studies reported that substantial amount of people indicates a willingness to use digital intervention, face-to-face psychotherapy, still, appeared to be the more preferred option(Renn et al., 2019). Thus, more research is needed to ascertain why people with depressive symptoms maintained a preference for in-person psychotherapy as opposed to the equally effective (Andersson, Titov, Dear, Rozental, &Carlbring, 2019) and yet cheaper options in digital form(Axelsson, Andersson, Ljótsson, &Hedman-Lagerlöf, 2018), and to examine what determinants facilitate its acceptance. Nevertheless, most of the current evidence on E-preference and acceptability were based on community sample. Not using samples with depressive symptoms above clinical threshold may limit the ecological validity of any conclusions drawn, as participants had to "imagine" whether they would use the services if they were undergoing a depressive episode, which could be cognitively demanding.

In fact, integration of digital treatment into health care systems is no small investment, especially when advanced techniques in computational and data science are increasingly incorporated in the development of the E-treatments(Chien et al., 2020). It is thus worthwhile to study both the "within" treatment determinant of E-service acceptance, and "between" treatment determinants of E-service as a preferred option so as to facilitate dissemination in real world setting. Understanding the "within" treatment determinants could help us formulate general direction in marketing E-mental health service for those who are in contemplation of trying E-mental health, while understanding the "between" treatment determinant could inform our direction in direct-to-consumer marketing or social campaigns (Baumeister et al., 2014) that aim at increasing the market share of E-mental health services by convincing traditional service preferers to use E-mental health services. Eventually, with more potential service users who are flexible in treatment modality, or prefer E-service, facilitation of dissemination of E-mental health service could be achieved by creating increased "pull demand", such that demand are created from consumers and to be responded by clinical providers, decision makers or stakeholders(Santucci, McHugh, &Barlow, 2012).

Apart from the readiness for E-mental health among the general population, it is also important to understand if the population who are "hard to reach" are also ready for E-mental health service, given digital mental health interventions are often suggested to be able to increase reach and access to special groups who may less well served by traditional mental health services (for example, people with financial difficulties(Andrade et al., 2014), men with depression or endorse masculinity norm(Seidler, Dawes, Rice, Oliffe, &Dhillon, 2016), and people with high level of stigma(Clement et al., 2015)). It is often assumed that E-mental health interventions are associated with a number of benefits over traditional face-to-face care(P.Musiat &Tarrier, 2014). While it may be theoretically true that e-mental health interventions increased anonymity, increased convenience with regards to time and location of treatment, reduced treatment cost and certain attitudinal barriers (Andersson et al., 2019; Spurgeon &Wright, 2010), it is unclear whether these "added benefits" enable individuals carrying the "hard to reach" characteristics prefer or accept E-service. It has also been suggested that the current evidence base for these "collateral outcomes" is sparse (P.Musiat &Tarrier, 2014), and the benefit of digital health interventions should be based on evidence, otherwise the "hard to reach" may left unreached when they are assumed to be reached by digital health interventions.

1.2 The applicability of Decision Aids (DAs) in clarify preference of psychotherapies Another important and yet unexplored issue on clients' preference of E-mental health service for depression is the applicability of Decision Aids (DAs). Making decision of health management, especially a preference sensitive one, requires skills. Decision makers of health services first need to acquire information of available option, then they have to identify, understand, and evaluate the options, and finally they need to select the best option with the consideration of personal situations and values. In the last decade, active participation of clients and patients in the decision making process regarding their health care has been increasingly advocated(Berry, Beckham, Dettman, &Mead, 2014). One of the influential conceptual models proposed within client-centered perspective of health care is the shared decision-making model. Shared decision-making model is a process of joint deliberation and collaboration between the health service providers and the clients in order to reach a consensus about treatment decisions. In this dyadic interaction, health service providers offer technical information about the disease or health condition, the benefits, and risks of the available therapeutic options, whereas the clients or patients provide information about their beliefs, concerns, values, and preferences about the consequences of those options(Joseph-Williams, Elwyn, &Edwards, 2014). Shared decision-making model is especially relevant when evidence indicated that available treatments showed a similar balance between benefits and risks, and when there is potential trade-off between different attributes of treatment options. In light of the above model, patients decision aids (DAs) are designed to promote and facilitate shared decision-making and help clients to make informed choices(Coulter et al., 2013). These materials are developed in different formats (e.g., paper and pen instruments, videos, audio, website and interactive software), and can be used alone by the client or in interaction with the health service providers. DAs include explanations about treatment options, describing the benefits and harms based on the scientific evidence, and characteristics of health service based on local situations. They also encourage patients to think about their own values and preferences regarding the benefits, risks, and different aspects of the different treatment options, and how the choices could influence their lives and well-being(Fagerlin et al., 2013). Recent systematic reviews show that DAs are effective in improving patients' knowledge about available treatments, and reduced decisional conflict (i.e., uncertainty about the course of action to take). They also have shown to reduce the proportion of people who were passive and undecisive in decision making after deliberation(Stacey et al., 2017).

In the specific area of depressive disorders, results show that a majority of people with depression are interested in receiving information about their illness and participating in shared and informed decision making(Loh et al., 2004; Perestelo-Perez et al., 2017). Unfortunately, studies found that people with depression often perceived a lesser involvement in decisions than they desire (Delas Cuevas, Peñate, &deRivera, 2014; Patel &Bakken, 2010). Moreover, despite this unmet demand, and while DAs had been widely and successfully adopted in the multiple arenas of physical health (such as, breast cancer treatment(Savelberg et al., 2017), HIV preexposure prophylaxis(Sewell et al., 2021), colon cancer screening(Miller et al., 2011)(see figure 1), and smoking cessation(Gültzow, Smit, Hudales, Dirksen, &Hoving, 2020)), there have been very few studies that have assessed the effectiveness of DAs in the field of depressive disorders. To our best knowledge no study has included E-mental health service in DAs for depression even when psychotherapy in E-format had been recommended by NICE for over a decade(Nice, 2009), and the effects of DAs on preference of psychological treatments and decisional conflict remain largely unknown.

1.3 Study Goal and Objective The goal of this study is to examine whether treatment preferences shift after receiving a clients' decision aids about psychotherapy in digital and in in-person format.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older;
* With at least mild to moderate depressive symptoms (defined as having a cut-off score of 10 or above based on the PHQ-9, Patient Health Questionnaire-9)
* Being Chinese speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2022-03-20 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Decisional conflict | Immediately before and right after (within 10 mins) the completion of the intervention.
  The decisional conflict scale (DCS) SURE-test

SECONDARY OUTCOMES:
Stage of decision making | Immediately before and right after (within 10 mins) the completion of the intervention.
  The Stage of Decision Making Scale measures individuals' readiness to engage in decision-making. It consists of a single item with six response options from 'haven't started to think about the choices' to 'have already made a decision and am unlikely to change my mind'. Earlier stages of decision-making are associated with higher levels of decisional conflict and vice versa.
Satisfaction with Decision (SWD) Scale | Immediately before and right after (within 10 mins) the completion of the intervention.
  SWD is a six-item Likert scale rated from 1= "strongly disagree" to 5 = "strongly agree" to assess satisfaction with the decision, with higher scores indicating higher levels of satisfaction. Sample items include "I am satisfied that I am adequately informed about the issues important to my decision."
Perceived benefits and risks | Immediately before and right after (within 10 mins) the completion of the intervention.
  Participants were asked to rate the degree to which they perceived face-to-face psychotherapy and guided Internet-based psychological intervention to be effective by indicating their estimation of the proportion of people with depression has clinically significant improvement on depressive symptoms after receiving the corresponding services from 0-100%, and their estimation of the proportion of people with depression has negative effect on depressive symptoms after receiving the corresponding services from 0-100%.
Service Preference Identity | Immediately before and right after (within 10 mins) the completion of the intervention.
  Two items were used to assess participants' service preference identity, with one item assessing personal liking, and the other item assessing likelihood of use. Participants were asked to indicate their preference (liking/favour) for either traditional face-to-face or guided Internet-based psychological intervention as their "preferred treatment option." An "unsure" option was included. Participants who chose guided Internet-based psychological intervention in this item were classified as "e-preferer." Then, participants were asked to indicate their preference between traditional face-to-face psychotherapy or guided Internet-based psychological intervention as a treatment option they would "likely to use." Again, an "unsure" option was included. Participants who selected guided Internet-based psychological intervention in this item were classified as "e-service inclined individuals."

OTHER OUTCOMES:
Depressive symtoms | Before intervention
  Depression severity was measured by the PHQ-9 (Patient Health Questionaire), which provides a brief measure of current depression symptoms using a 4-point Likert scale ranging from 0 (not at all) to 3 (nearly every day) in the past 2 weeks. The minimum and maximum values are 0 and 27, with higher score indicate higher depressive symtpoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychology, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Practice guideline for the treatment of patients with major depressive disorder (revision). American Psychiatric Association. Am J Psychiatry. 2000 Apr;157(4 Suppl):1-45. No abstract available. PMID 10767867
- [Background] Andersson G, Titov N, Dear BF, Rozental A, Carlbring P. Internet-delivered psychological treatments: from innovation to implementation. World Psychiatry. 2019 Feb;18(1):20-28. doi: 10.1002/wps.20610. PMID 30600624
- [Background] Andrade LH, Alonso J, Mneimneh Z, Wells JE, Al-Hamzawi A, Borges G, Bromet E, Bruffaerts R, de Girolamo G, de Graaf R, Florescu S, Gureje O, Hinkov HR, Hu C, Huang Y, Hwang I, Jin R, Karam EG, Kovess-Masfety V, Levinson D, Matschinger H, O'Neill S, Posada-Villa J, Sagar R, Sampson NA, Sasu C, Stein DJ, Takeshima T, Viana MC, Xavier M, Kessler RC. Barriers to mental health treatment: results from the WHO World Mental Health surveys. Psychol Med. 2014 Apr;44(6):1303-17. doi: 10.1017/S0033291713001943. Epub 2013 Aug 9. PMID 23931656
- [Background] Angermeyer MC, Matschinger H, Riedel-Heller SG. Whom to ask for help in case of a mental disorder? Preferences of the lay public. Soc Psychiatry Psychiatr Epidemiol. 1999 Apr;34(4):202-10. doi: 10.1007/s001270050134. PMID 10365626
- [Background] Axelsson E, Andersson E, Ljotsson B, Hedman-Lagerlof E. Cost-effectiveness and long-term follow-up of three forms of minimal-contact cognitive behaviour therapy for severe health anxiety: Results from a randomised controlled trial. Behav Res Ther. 2018 Aug;107:95-105. doi: 10.1016/j.brat.2018.06.002. Epub 2018 Jun 15. PMID 29936239
- [Background] Baumeister H, Nowoczin L, Lin J, Seifferth H, Seufert J, Laubner K, Ebert DD. Impact of an acceptance facilitating intervention on diabetes patients' acceptance of Internet-based interventions for depression: a randomized controlled trial. Diabetes Res Clin Pract. 2014 Jul;105(1):30-9. doi: 10.1016/j.diabres.2014.04.031. Epub 2014 May 10. PMID 24862240
- [Background] Berry LL, Beckham D, Dettman A, Mead R. Toward a strategy of patient-centered access to primary care. Mayo Clin Proc. 2014 Oct;89(10):1406-15. doi: 10.1016/j.mayocp.2014.06.011. Epub 2014 Sep 4. PMID 25199953
- [Background] Carlbring P, Andersson G, Cuijpers P, Riper H, Hedman-Lagerlof E. Internet-based vs. face-to-face cognitive behavior therapy for psychiatric and somatic disorders: an updated systematic review and meta-analysis. Cogn Behav Ther. 2018 Jan;47(1):1-18. doi: 10.1080/16506073.2017.1401115. Epub 2017 Dec 7. PMID 29215315
- [Background] Cavanagh K, Shapiro DA, Van Den Berg S, Swain S, Barkham M, Proudfoot J. The acceptability of computer-aided cognitive behavioural therapy: a pragmatic study. Cogn Behav Ther. 2009;38(4):235-46. doi: 10.1080/16506070802561256. PMID 19306147
- [Background] Chien I, Enrique A, Palacios J, Regan T, Keegan D, Carter D, Tschiatschek S, Nori A, Thieme A, Richards D, Doherty G, Belgrave D. A Machine Learning Approach to Understanding Patterns of Engagement With Internet-Delivered Mental Health Interventions. JAMA Netw Open. 2020 Jul 1;3(7):e2010791. doi: 10.1001/jamanetworkopen.2020.10791. PMID 32678450
- [Background] Clement S, Brohan E, Jeffery D, Henderson C, Hatch SL, Thornicroft G. Development and psychometric properties the Barriers to Access to Care Evaluation scale (BACE) related to people with mental ill health. BMC Psychiatry. 2012 Jun 20;12:36. doi: 10.1186/1471-244X-12-36. PMID 22546012
- [Background] Clement S, Schauman O, Graham T, Maggioni F, Evans-Lacko S, Bezborodovs N, Morgan C, Rusch N, Brown JS, Thornicroft G. What is the impact of mental health-related stigma on help-seeking? A systematic review of quantitative and qualitative studies. Psychol Med. 2015 Jan;45(1):11-27. doi: 10.1017/S0033291714000129. Epub 2014 Feb 26. PMID 24569086
- [Background] Coulter A, Stilwell D, Kryworuchko J, Mullen PD, Ng CJ, van der Weijden T. A systematic development process for patient decision aids. BMC Med Inform Decis Mak. 2013;13 Suppl 2(Suppl 2):S2. doi: 10.1186/1472-6947-13-S2-S2. Epub 2013 Nov 29. PMID 24625093
- [Background] Cuijpers P, Clignet F, van Meijel B, van Straten A, Li J, Andersson G. Psychological treatment of depression in inpatients: a systematic review and meta-analysis. Clin Psychol Rev. 2011 Apr;31(3):353-60. doi: 10.1016/j.cpr.2011.01.002. Epub 2011 Jan 16. PMID 21382540
- [Background] De las Cuevas C, Penate W, de Rivera L. Psychiatric patients' preferences and experiences in clinical decision-making: examining concordance and correlates of patients' preferences. Patient Educ Couns. 2014 Aug;96(2):222-8. doi: 10.1016/j.pec.2014.05.009. Epub 2014 May 22. PMID 24894880
- [Background] Lubas B, Wilczok T. Spin-echo technique study of the non-rotational hydration of deoxyribonucleic acid. Biochim Biophys Acta. 1966 Jul 13;120(3):427-33. doi: 10.1016/0926-6585(66)90309-8. No abstract available. PMID 5966543
- [Background] Witteman HO, Ndjaboue R, Vaisson G, Dansokho SC, Arnold B, Bridges JFP, Comeau S, Fagerlin A, Gavaruzzi T, Marcoux M, Pieterse A, Pignone M, Provencher T, Racine C, Regier D, Rochefort-Brihay C, Thokala P, Weernink M, White DB, Wills CE, Jansen J. Clarifying Values: An Updated and Expanded Systematic Review and Meta-Analysis. Med Decis Making. 2021 Oct;41(7):801-820. doi: 10.1177/0272989X211037946. PMID 34565196
- [Background] Gelhorn HL, Sexton CC, Classi PM. Patient preferences for treatment of major depressive disorder and the impact on health outcomes: a systematic review. Prim Care Companion CNS Disord. 2011;13(5):PCC.11r01161. doi: 10.4088/PCC.11r01161. PMID 22295273
- [Background] Harter M, Klesse C, Bermejo I, Bschor T, Gensichen J, Harfst T, Hautzinger M, Kolada C, Kopp I, Kuhner C, Lelgemann M, Matzat J, Meyerrose B, Mundt C, Niebling W, Ollenschlager G, Richter R, Schauenburg H, Schulz H, Weinbrenner S, Schneider F, Berger M. [Evidence-based therapy of depression: S3 guidelines on unipolar depression]. Nervenarzt. 2010 Sep;81(9):1049-68. doi: 10.1007/s00115-010-3084-7. German. PMID 20802992
- [Background] Givens JL, Houston TK, Van Voorhees BW, Ford DE, Cooper LA. Ethnicity and preferences for depression treatment. Gen Hosp Psychiatry. 2007 May-Jun;29(3):182-91. doi: 10.1016/j.genhosppsych.2006.11.002. PMID 17484934
- [Background] Gultzow T, Smit ES, Hudales R, Dirksen CD, Hoving C. Smoker profiles and their influence on smokers' intention to use a digital decision aid aimed at the uptake of evidence-based smoking cessation tools: An explorative study. Digit Health. 2020 Dec 29;6:2055207620980241. doi: 10.1177/2055207620980241. eCollection 2020 Jan-Dec. PMID 33473322
- [Background] Hanson K, Webb TL, Sheeran P, Turpin G. Attitudes and Preferences towards Self-help Treatments for Depression in Comparison to Psychotherapy and Antidepressant Medication. Behav Cogn Psychother. 2016 Mar;44(2):129-39. doi: 10.1017/S1352465815000041. Epub 2015 Feb 20. PMID 25697236
- [Background] Hockenberry JM, Joski P, Yarbrough C, Druss BG. Trends in Treatment and Spending for Patients Receiving Outpatient Treatment of Depression in the United States, 1998-2015. JAMA Psychiatry. 2019 Aug 1;76(8):810-817. doi: 10.1001/jamapsychiatry.2019.0633. PMID 31017627
- [Background] Joseph-Williams N, Elwyn G, Edwards A. Knowledge is not power for patients: a systematic review and thematic synthesis of patient-reported barriers and facilitators to shared decision making. Patient Educ Couns. 2014 Mar;94(3):291-309. doi: 10.1016/j.pec.2013.10.031. Epub 2013 Nov 9. PMID 24305642
- [Background] Josephine K, Josefine L, Philipp D, David E, Harald B. Internet- and mobile-based depression interventions for people with diagnosed depression: A systematic review and meta-analysis. J Affect Disord. 2017 Dec 1;223:28-40. doi: 10.1016/j.jad.2017.07.021. Epub 2017 Jul 10. PMID 28715726
- [Background] Kaltenthaler E, Sutcliffe P, Parry G, Beverley C, Rees A, Ferriter M. The acceptability to patients of computerized cognitive behaviour therapy for depression: a systematic review. Psychol Med. 2008 Nov;38(11):1521-30. doi: 10.1017/S0033291707002607. Epub 2008 Jan 21. PMID 18205964
- [Background] Kenwright M, Marks I, Gega L, Mataix-Cols D. Computer-aided self-help for phobia/panic via internet at home: a pilot study. Br J Psychiatry. 2004 May;184:448-9. doi: 10.1192/bjp.184.5.448. PMID 15123511
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Loh A, Kremer N, Giersdorf N, Jahn H, Hanselmann S, Bermejo I, Harter M. [Information and participation interests of patients with depression in clinical decision making in primary care]. Z Arztl Fortbild Qualitatssich. 2004 Mar;98(2):101-7. German. PMID 15106488
- [Background] Mahoney A, Li I, Haskelberg H, Millard M, Newby JM. The uptake and effectiveness of online cognitive behaviour therapy for symptoms of anxiety and depression during COVID-19. J Affect Disord. 2021 Sep 1;292:197-203. doi: 10.1016/j.jad.2021.05.116. Epub 2021 Jun 4. PMID 34126311
- [Background] March S, Day J, Ritchie G, Rowe A, Gough J, Hall T, Yuen CYJ, Donovan CL, Ireland M. Attitudes Toward e-Mental Health Services in a Community Sample of Adults: Online Survey. J Med Internet Res. 2018 Feb 19;20(2):e59. doi: 10.2196/jmir.9109. PMID 29459357
- [Background] McCall HC, Sison AP, Burnett JL, Beahm JD, Hadjistavropoulos HD. Exploring Perceptions of Internet-Delivered Cognitive Behaviour Therapy among Public Safety Personnel: Informing Dissemination Efforts. Int J Environ Res Public Health. 2020 Aug 19;17(17):6026. doi: 10.3390/ijerph17176026. PMID 32824994
- [Background] von Kleist S. The clinical value of the tumor markers CA 19/9 and carcinoembryonic antigen (CEA) in colorectal carcinomas: a critical comparison. Int J Biol Markers. 1986 Jan-Apr;1(1):3-8. doi: 10.1177/172460088600100102. PMID 3480321
- [Background] Murray CJ, Lopez AD. Measuring the global burden of disease. N Engl J Med. 2013 Aug 1;369(5):448-57. doi: 10.1056/NEJMra1201534. No abstract available. PMID 23902484
- [Background] Musiat P, Goldstone P, Tarrier N. Understanding the acceptability of e-mental health--attitudes and expectations towards computerised self-help treatments for mental health problems. BMC Psychiatry. 2014 Apr 11;14:109. doi: 10.1186/1471-244X-14-109. PMID 24725765
- [Background] Musiat P, Tarrier N. Collateral outcomes in e-mental health: a systematic review of the evidence for added benefits of computerized cognitive behavior therapy interventions for mental health. Psychol Med. 2014 Nov;44(15):3137-50. doi: 10.1017/S0033291714000245. Epub 2014 Feb 19. PMID 25065947
- [Background] National Collaborating Centre for Mental Health (UK). Depression: The Treatment and Management of Depression in Adults (Updated Edition). Leicester (UK): British Psychological Society; 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK63748/ PMID 22132433
- [Background] O'Connor AM. Validation of a decisional conflict scale. Med Decis Making. 1995 Jan-Mar;15(1):25-30. doi: 10.1177/0272989X9501500105. PMID 7898294
- [Background] Stacey D, Legare F, Boland L, Lewis KB, Loiselle MC, Hoefel L, Garvelink M, O'Connor A. 20th Anniversary Ottawa Decision Support Framework: Part 3 Overview of Systematic Reviews and Updated Framework. Med Decis Making. 2020 Apr;40(3):379-398. doi: 10.1177/0272989X20911870. PMID 32428429
- [Background] Patel SR, Bakken S. Preferences for participation in decision making among ethnically diverse patients with anxiety and depression. Community Ment Health J. 2010 Oct;46(5):466-73. doi: 10.1007/s10597-010-9323-3. Epub 2010 Jun 17. PMID 20556512
- [Background] Perestelo-Perez L, Rivero-Santana A, Sanchez-Afonso JA, Perez-Ramos J, Castellano-Fuentes CL, Sepucha K, Serrano-Aguilar P. Effectiveness of a decision aid for patients with depression: A randomized controlled trial. Health Expect. 2017 Oct;20(5):1096-1105. doi: 10.1111/hex.12553. Epub 2017 Mar 10. PMID 28295915
- [Background] Rahimi AR, Spertus JA, Reid KJ, Bernheim SM, Krumholz HM. Financial barriers to health care and outcomes after acute myocardial infarction. JAMA. 2007 Mar 14;297(10):1063-72. doi: 10.1001/jama.297.10.1063. PMID 17356027
- [Background] Raue PJ, Schulberg HC, Heo M, Klimstra S, Bruce ML. Patients' depression treatment preferences and initiation, adherence, and outcome: a randomized primary care study. Psychiatr Serv. 2009 Mar;60(3):337-43. doi: 10.1176/ps.2009.60.3.337. PMID 19252046
- [Background] Renn BN, Hoeft TJ, Lee HS, Bauer AM, Arean PA. Preference for in-person psychotherapy versus digital psychotherapy options for depression: survey of adults in the U.S. NPJ Digit Med. 2019 Feb 11;2:6. doi: 10.1038/s41746-019-0077-1. eCollection 2019. PMID 31304356
- [Background] Santucci LC, McHugh RK, Barlow DH. Direct-to-consumer marketing of evidence-based psychological interventions: introduction. Behav Ther. 2012 Jun;43(2):231-5. doi: 10.1016/j.beth.2011.07.003. Epub 2011 Jul 28. PMID 22440061
- [Background] Savelberg W, van der Weijden T, Boersma L, Smidt M, Willekens C, Moser A. Developing a patient decision aid for the treatment of women with early stage breast cancer: the struggle between simplicity and complexity. BMC Med Inform Decis Mak. 2017 Aug 1;17(1):112. doi: 10.1186/s12911-017-0505-6. PMID 28764688
- [Background] Seidler ZE, Dawes AJ, Rice SM, Oliffe JL, Dhillon HM. The role of masculinity in men's help-seeking for depression: A systematic review. Clin Psychol Rev. 2016 Nov;49:106-118. doi: 10.1016/j.cpr.2016.09.002. Epub 2016 Sep 10. PMID 27664823
- [Background] Sewell WC, Solleveld P, Seidman D, Dehlendorf C, Marcus JL, Krakower DS. Patient-Led Decision-Making for HIV Preexposure Prophylaxis. Curr HIV/AIDS Rep. 2021 Feb;18(1):48-56. doi: 10.1007/s11904-020-00535-w. Epub 2021 Jan 8. PMID 33417201
- [Background] Spurgeon JA, Wright JH. Computer-assisted cognitive-behavioral therapy. Curr Psychiatry Rep. 2010 Dec;12(6):547-52. doi: 10.1007/s11920-010-0152-4. PMID 20872100
- [Background] Stacey D, Legare F, Lewis K, Barry MJ, Bennett CL, Eden KB, Holmes-Rovner M, Llewellyn-Thomas H, Lyddiatt A, Thomson R, Trevena L. Decision aids for people facing health treatment or screening decisions. Cochrane Database Syst Rev. 2017 Apr 12;4(4):CD001431. doi: 10.1002/14651858.CD001431.pub5. PMID 28402085
- [Background] Steidtmann D, Manber R, Arnow BA, Klein DN, Markowitz JC, Rothbaum BO, Thase ME, Kocsis JH. Patient treatment preference as a predictor of response and attrition in treatment for chronic depression. Depress Anxiety. 2012 Oct;29(10):896-905. doi: 10.1002/da.21977. Epub 2012 Jul 5. PMID 22767424
- [Background] Swift JK, Callahan JL. The impact of client treatment preferences on outcome: a meta-analysis. J Clin Psychol. 2009 Apr;65(4):368-81. doi: 10.1002/jclp.20553. PMID 19226606
- [Background] Taylor S, Landry CA, Paluszek MM, Fergus TA, McKay D, Asmundson GJG. Development and initial validation of the COVID Stress Scales. J Anxiety Disord. 2020 May;72:102232. doi: 10.1016/j.janxdis.2020.102232. Epub 2020 May 4. PMID 32408047
- [Background] Wallin EE, Mattsson S, Olsson EM. The Preference for Internet-Based Psychological Interventions by Individuals Without Past or Current Use of Mental Health Treatment Delivered Online: A Survey Study With Mixed-Methods Analysis. JMIR Ment Health. 2016 Jun 14;3(2):e25. doi: 10.2196/mental.5324. PMID 27302200
- [Background] Wills CE, Holmes-Rovner M. Preliminary validation of the Satisfaction With Decision scale with depressed primary care patients. Health Expect. 2003 Jun;6(2):149-59. doi: 10.1046/j.1369-6513.2003.00220.x. PMID 12752743
- [Derived] Auyeung L, Mak WW, Tsang EZ, Yang PL. Impact of a Digital Decision Aid When Choosing Between Face-to-Face and Guided Internet-Based Psychological Interventions for Depression Among Chinese-Speaking Participants in Hong Kong: Randomized Controlled Trial. J Med Internet Res. 2025 May 6;27:e54727. doi: 10.2196/54727. PMID 40327376